CLINICAL TRIAL: NCT04240600
Title: Effect of a Hyperproteic Hyperenergetic Enteral Formula on Body Composition, Muscle Strength and Concentration of Vascular Endothelial Growth Factor (VEGF) in Patients With Actue Myeloid Leukemia (AML) During the Hospital Stay
Brief Title: Effect of a Hyperproteic Hyperenergetic Enteral Formula on Body Composition and VEGF in AML During Hospital Stay
Acronym: HEMVEF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General de Mexico (Other Government)
Collaborators: Fresenius Kabi (Industry)
Responsible Party: Principal Investigator, Dr. Vanessa Fuchs Tarlovsky, Principal Investigator, Hospital General de Mexico
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DI/19/11/03/017
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Acute Myeloid Leukemia, Adult
Keywords: nutrition; acute myeloid leukemia; body composition; chemotherapy recovery; VEGF
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: A randomized clinical trial study
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hyperproteic, hypercaloric formula (Experimental): Each patient will receive 2 bottles per day of Supportan DKN during the hospital stay (nutritional contribution: 600 kcal and 40 g of protein).
  Interventions: Dietary Supplement: Experimental group
- Standard formula (Active Comparator): Each patient will receive 2 cans or bottles per day of Fresubin® Original DRINK (nutritional contribution: 474.2 kcal and 17.6 g of protein).
  Interventions: Dietary Supplement: Control group

INTERVENTIONS:
Dietary Supplement: Experimental group — 2 cans or bottles (200ml)per day, orally
  Other Names: Supportan DKN
  Arms: Hyperproteic, hypercaloric formula
Dietary Supplement: Control group — 2 cans or bottles (200ml)per day, orally
  Other Names: Fresubin® Original DRINK
  Arms: Standard formula

SUMMARY:
A randomized controlled clinical trial in two groups of supplementation with high protein enteral formula and a normocaloric enteral formula in two groups of 37 patients .

DETAILED DESCRIPTION:
Patients with acute myeloid leukemia have a high risk of suffering sarcopenia, which decreases the oncology therapy clinical response, functional ability and quality of life. Chemotherapy is used in these patients, some of them inhibit angiogenesis and act in an important way in physiological processes of muscle anabolism. The vascular endothelial growth factor (VEGF) and its receptors (VEGFR) play a crucial role in both normal and malignant angiogenesis. Activation of the VEGF pathway leads to endothelial cell activation, proliferation and survival.

The objective of this study is to compare the effect of the use of a high protein, high energy enteral with omega 3 formula (Supportan DKN) against a standard enteral formula (Fresubin® Original DRINK) on body composition, days of hospital stay, quality of life, associated muscular strength with levels of VEGF in patients with acute myeloid leukemia during induction chemotherapy.

An open clinical trial was designed, in which a group of patients will receive, as part of their nutritional requirements a hyperproteic hyperenergetic enteral formula versus standard formula during the 21 days of the first cycle of antineoplastic treatment. We will measure body composition, muscle strength and serum concentrations of VEGFR in both groups to be able to compare its effect.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with a confirmed diagnosis of AML
* Tolerance to oral feeding
* Induction Chemotherapy
* Patients with nutritional risk of positive malnutrition (Score +3 NRS).
* Candidates to receive enteral nutrition, as well as chemotherapy according to medical indications.
* Life expectancy greater than a week and with the possibility of starting oncological treatment. Have informed consent obtained by the patient prior to randomization

Exclusion Criteria:

* Geriatric patients (> 60 years)
* Patients with acute gastrointestinal bleeding, ileus and shock
* History of recurrence of neoplasm
* Renal failure
* Atrophy of the gastrointestinal mucosa
* Central nervous system disease,
* impaired cardiac function.

Elimination criteria:

Lack of follow up Incomplete data. Insufficient amount of genetic material to perform the determination of the VEGF material.

Absence of the determination of the levels of VEGF prior to the start of oncological therapy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2020-12-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Effect of use of hyperproteic, hypercaloric enteral formula in body composition and VEGF | 21 days
  The aim of this study is to compare the effect of the use of a hyperproteic hypercaloric enteral formula (Supportan DKN.) With a standard enteral formula (Fresubin® Original DRINK) in patients with AML during antineoplastic treatment.

SECONDARY OUTCOMES:
Body composition fat mass | 21 days
  To messured fat mass with seca mBCA 525medical Body Composition Analyzer at the beginning and after intervention therapy.
Body compositition: fat-free mass | 21 days
  To messured fat-free mass with seca mBCA 525medical Body Composition Analyzer at the beginning and after intervention therapy.
Body composition: phase angle | 21 days
  To messured phase angle with seca mBCA 525medical Body Composition Analyzer at the beginning and after intervention therapy.
SARC-F | 21 days
  To evaluate the score of SARC-F (an scale of symptoms to predict patients with sarcopenia at risk of low functional outcome) at the beginning and after intervention therapy.
Length of stay | It depends of the patients health condition
  To evaluate the length of stay (in days) of their induction chemotherapy recovery
Early mortality | 21 days
  Estimation of early mortality (first three weeks) in patients receiving chemotherapy treatment
Late mortality | 1 year
  Estimation of late mortality (one-year follow-up) in patients receiving chemotherapy
Changes in nutritional status during oncological therapy | 21 days
  To documented in text format presence of changes in nutritional status according biochemical,clinical and anthropometric paramethers . This changes will be evaluated by a standarized nutricionist acording ESPEN guideliness for oncological patients
Evaluation of the quality of life at the beginning and after the intervention. | 21 days
  To evaluate the score of the European Organization for Research and Treatment of Cancer (EORTC) at the beginning and after intervention therapy.
Levels of VEGF | 2 years
  To determinate cuantitative levels of VEGF´s RNA expression at the beginning and after treatment
Response to induction chemotherapy. | 28 days
  To evaluate response to induction chemotherapy from to blast citometry percentaje
Early biochemical recovery values | 28 days
  To evaluate the recovery of platelets, neutrophils, hemoglobin

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Fuchs Tarlovsky, PhD, Study Director — Hospital General de México
Locations (2):
- Mexico (2):
  - Vannesa Fuchs Tarlovsky, Mexico City
  - Hospital General de México, Mexico City